CLINICAL TRIAL: NCT06398314
Title: Palliative Radiotherapy in Symptomatic Pelvic Soft Tissue Tumors
Acronym: PALLSOFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Telemark (Other Government)
Collaborators: Nordlandssykehuset HF (Other); Møre og Romsdal Hospital Trust (Other); Helse Stavanger HF (Other Government); Hospital of Southern Norway Trust (Other); Oslo University Hospital (Other); Vestre Viken Hospital Trust (Other); Sykehuset Innlandet HF (Other); St. Olavs Hospital (Other); Haukeland University Hospital (Other); University Hospital of North Norway (Other); South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 606316 (REK)
Record Dates: First submitted 2024-04-17; First posted 2024-05-03 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-03

CONDITIONS: Gastrointestinal Cancer; Urologic Cancer; Gynecologic Cancer
Keywords: Palliative radiotherapy; Patient-reported outcomes; Gastrointestinal cancer; Urologic cancer; Gynecologic cancer; Tumor hypoxia
MeSH Terms: conditions — Gastrointestinal Neoplasms; Urologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Non-inferiority, multicenter
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1-2 fractions of 8 Gy (Gray) (Active Comparator)
  Interventions: Radiation: Palliative radiotherapy
- 5 fractions of 5 Gy (Gray) (Active Comparator)
  Interventions: Radiation: Palliative radiotherapy

INTERVENTIONS:
Radiation: Palliative radiotherapy — Hypofractionated radiotherapy

SUMMARY:
PALLSOFT is a randomized, open-label, non-inferiority phase III, multicenter, national trial that will investigate whether the patient-reported symptomatic effect of palliative radiotherapy delivered in 1-2 fractions is non-inferior to palliative radiotherapy delivered in five fractions in patients with pelvic soft tissue tumors from either gastrointestinal, urological or gynecological cancer. Health-related quality of life, toxicities, survival and prognostic and predictive biomarkers will be assessed as secondary and explorative endpoints.

DETAILED DESCRIPTION:
Studies and clinical practice have proven palliative radiotherapy to provide efficient symptom relief in patients with symptomatic pelvic soft tissue tumors. However, studies are mainly retrospective, are difficult to compare due to a variety of radiotherapy fractionation schedules used, and lack data on patient-reported quality of life. Consequently, no recommended standard of care is established, and several schedules are employed with variations in both number of fractions and total radiation dose (measured in Gray=Gy). Given the limited life expectancy of palliative patients, a short-course radiotherapy schedule would be preferable provided efficient symptom relief and good health-related quality of life.

PALLSOFT is a national, randomized, non-inferiority study that will investigate whether the symptomatic effect of a short-course radiotherapy schedule of 8 Gy x 1-2 is non-inferior to a more prolonged schedule of 5 Gy x 5. The study will include patients with symptomatic pelvic soft tissue tumors from either gastrointestinal, urological or gynecological cancer. Patients will defined a target symptom from 5 predefined cathegories (pain, bleeding, bowel/lower urinary tract/vaginal dysfunction), and change in symptom intensity will be assessed, as well as overall toxicities, quality of life and survival. Prognostic and predictive biomarkers will be explores, the latter with particular emphasis on the significance of tumor hypoxia in palliative radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients unsuitable for curative treatment due to either advanced disease or medical contradictions (i.e comorbidity, old age, poor general condition)
* Histologically verified primary cancer originated from gastrointestinal, urological or gynecological organs (histological verification can be performed on other lesions than the symptomatic pelvic tumor)
* Primary, residual, recurrent or metastatic pelvic tumor from the above-mentioned cancers not amenable for curative treatment
* Tumor-related symptoms including within the 5 defined categories pain, bleeding, bowel/lower urinary/vaginal dysfunction
* Considered candidate for palliative radiotherapy according to both study arms
* Patient reported severity of symptoms ≥4 on a NRS- scale of 0-10
* ≥18 years of age
* Speaks and understands Norwegian or English
* Ability to understand and willing to sign a written informed consent
* ECOG performance status 0-3
* Expected survival > 12 weeks
* Able to pause systemic cancer treatment for one week prior to, during, and one week after the radiotherapy treatment
* Women of childbearing potential (WOCBP) should have a negative highly sensitive serum pregnancy test within 72 hours prior to study intervention. WOCBP must agree to the use of highly effective birth control methods or abstain from heterosexual sexual activity from randomization and until completed study intervention

Exclusion Criteria:

* Neuroendocrine histology of any kind
* Sarcoma or sarcomal components in the histology
* Tumors that originate from bony metastases without a soft tissue component
* Unable to comply with study questionnaires
* Ongoing treatment with an investigational drug at inclusion
* Planned inclusion in another interventional clinical trial within 4 weeks after radiotherapy
* Patients who are pregnant due to risk of teratogenic and abortifacient effects of radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Patient-reported symptomatic effect | 12 weeks
  Establish whether 1-2 fractions of 8 Gy is non-inferior to 5 fractions of 5 Gy with regards to target symptom effect assessed by change in NRS 0-10 (Numerical Rating Scale) from baseline

SECONDARY OUTCOMES:
Physician-reported toxicities | 52 weeks
  Establish whether 1-2 fractions of 8 Gy is non-inferior to 5 fractions of 5 Gy with regards to bladder and bowel toxicities assessed by CTCAE
Survival | 2 years
  Establish whether 1-2 fractions of 8 Gy is non-inferior to 5 fractions of 5 Gy with regards to overall survival

OTHER OUTCOMES:
Patient-reported quality of life | 12 weeks
  Establish whether 1-2 fractions of 8 Gy is non-inferior to 5 fractions of 5 Gy with regards to quality of life assessed by EORTC-QLQ C15PAL (European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core15 Palliative)
Prognostic models | Baseline
  Explore prognostic models for patient classification:
  Glasgow Prognostic Score (GPS): C-Reactive Protein (CRP, mg/L), Albumin (g/L) GPS 0 = Normal level CRP and albumin GPS 1: Increased CRP or low albumin GPS 2: Increased CRP and low albumin
Prognostic models | Baseline
  Explore prognostic models for patient classification:
  LabBM: CRP (mg/L), LDH (lactate dehydrogenase, U/L), Albumin (g/L), hemoglobin (g/dL), platelets (E09/L) The score is calculated as follows; CRP and LDH above upper limit of normal=1 point for each parameter. Albumin, hemoglobin and platelets below the lower limit of normal: 0.5 point for each parameter. Minimum score 0 point, maximum score 3.5 points. Low score indicates a more favorable prognosis
Prognostic models | Baseline
  Explore prognostic models for patient classification:
  LabPS: CRP (mg/L), LDH (lactate dehydrogenase, U/L), Albumin (g/L), hemoglobin (g/dL), platelets (E09/L), Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) The score is calculated as follows; CRP and LDH above upper limit of normal=1 point for each parameter. Albumin, hemoglobin and platelets below the lower limit of normal: 0.5 point for each parameter. ECOG PS 3-4, 2 and 0-1: 1, 0.5 and 0 points,respectively Minimum score 0 point, maximum score 4.5 points. Low score indicates a more favorable prognosis
Predictive biomarkers MRI | Baseline
  Magnetic Resonance Images (MRI) previously acquired for diagnosis, treatment and/or follow up will be collected. Hypoxia images will be generated using the Consumption and Supply- based Hypoxia (CSH) Imaging Method. The tumor hypoxic fraction (HF) will be calculated on hypoxia images and explored as a potential explanatory response variable in individual patients.
Predictive biomarkers tumor biopsies | Baseline
  Tumor biopsies previously acquired for diagnosis, treatment and/or follow up will be collected. Tumor RNA will be isolated from paraffin embedded tissue blocks, subjected to global gene expression analysis and used to indicate hypoxia by applying previously established gene signatures. Gene signatures will be explored as potential explanatory response variable in individual patients.

CONTACTS AND LOCATIONS:
Overall Officials: Harald Ragnum, MD,PhD, Study Chair — Telemark Hospital Trust
Locations (11):
- Norway (11):
  - Helse Møre og Romsdal, Ålesund
  - Haukeland universitetssykehus, Bergen
  - Nordlandssykehuset Bodø, Bodø
  - Vestre Viken HF, Drammen
  - Sykehuset Innlandet HF, Gjøvik
  - Sørlandet sykehus HF, Kristiansand
  - Oslo Universitetssykehus, Oslo
  - Sykehuset Telemark HF, Skien
  - Stavanger Universitetssykehus, Stavanger
  - Universitetssykehuset i Nord-Norge, Tromsø
  - St. Olavs Hospital HF, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Skipar K, Orvik MS, Evers C, Balteskard L, Ekanger C, Giske LE, Odegaard K, Ostrem EH, Nordstrand CS, Tondel H, Nieder C, Guren MG, Kaasa S, Ragnum HB. Palliative radiotherapy in symptomatic pelvic soft tissue tumors (PallSoft)- protocol for a national, randomized, non-inferiority study. BMC Cancer. 2025 Jul 1;25(1):1051. doi: 10.1186/s12885-025-14424-1. PMID 40597814